CLINICAL TRIAL: NCT01404364
Title: Use of Intravitreal Triamcinolone and Retrobulbar Chlorpromazine as Alternatives to the Management of Painful Blind Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Governador Celso Ramos (Other)
Responsible Party: Deborah Cristina Ribas, Hospital Governador Celso Ramos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HGCR-20101
Record Dates: First submitted 2011-07-11; First posted 2011-07-28 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Blind Painful Eye; Refractory Glaucoma; Control of Pain Through Drug Injection
Keywords: Triamcinolone; Chlorpromazine; Refractory glaucoma; Blind painful eye
MeSH Terms: conditions — Glaucoma | interventions — Triamcinolone; Chlorpromazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravitreal Triamcinolone (Active Comparator): Patients with phthisis bulbi received 0,3ml intravitreal triamcinolone injection
  Interventions: Drug: Triamcinolone
- Retrobulbar Chlorpromazine (Active Comparator): Patients with refractory glaucoma and blind painful eye were submitted to 2,5mL Chlorpromazine retrobulbar injection
  Interventions: Drug: Chlorpromazine

INTERVENTIONS:
Drug: Triamcinolone — 0,3mL intravitreal injection of Triamcinolone, single dose
  Arms: Intravitreal Triamcinolone
Drug: Chlorpromazine — 2,5mL Chlorpromazine retrobulbar injection, single dose
  Other Names: Amplictil
  Arms: Retrobulbar Chlorpromazine

SUMMARY:
The purpose of this study is to evaluate the efficacy of intravitreal triamcinolone and retrobulbar chlorpromazine as alternatives in the management of ocular pain in blind eyes.

DETAILED DESCRIPTION:
The management of chronic eye pain is a constant challenge to ophthalmology. Treatment varies with the intensity of pain, and topical eye drops and contact lens therapy are effective in many patients. In refractory cases, and without vision, surgical removal of the eye through enucleation is considered classical therapy. As less invasive alternatives we have cyclodestruction and neurolytic drug injection in order to promote analgesia for a prolonged period.

The purpose of this study is to evaluate the efficacy of intravitreal triamcinolone and retrobulbar chlorpromazine as alternatives in the management of This is a prospective study of patients with blind painful eyes not responsive to topical treatment and with no indication for evisceration seen at the Department of Ophthalmology, Hospital Governador Celso Ramos (HGCR) in 2010.

ELIGIBILITY:
Inclusion Criteria:

* patients treated in the period at HGCR who wanted to be part of the protocol by signing the consent form

Exclusion Criteria:

* patients whose follow-up period was less than three months

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in Pain intensity | 0, 1 month, 3 months, 6 months after procedure
  Pain was measured asking the patient to graduate it in a scale from 0 to 10, 0 being no pain, 10 being the worst pain patient has experienced in life

SECONDARY OUTCOMES:
Changes in Use of eyedrops before and after drug injection | 0, 1 month, 3 months, 6 months
  Patient use of eyedrops before and after the procedure (yes or no)
Changes in Intraocular pressure (IOP) | 0, 1 months, 3 months, 6 months
  IOP was measured at all times of patient evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Deborah C Ribas, MD, Principal Investigator — Hospital Governador Celso Ramos
Locations (1):
- Hospital Governador Celso Ramos, Florianópolis, Santa Catarina, Brazil